CLINICAL TRIAL: NCT00193115
Title: Phase II Pilot Trial of Dose-Dense Docetaxel Followed by Doxorubicin Plus Cyclophosphamide (T-AC) Given as Adjuvant or Neoadjuvant Treatment for Women With Node Positive or High-Risk Primary Breast Cancer
Brief Title: Docetaxel Followed by Doxorubicin Plus Cyclophosphamide for Node Positive or High-Risk Primary Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Denise A. Yardley, M.D., Sarah Cannon Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 69; 11251
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2009-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Doxorubicin; Cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel
Drug: Doxorubicin
Drug: Cyclophosphamide

SUMMARY:
This protocol will evaluate the feasibility and toxicity of dose-dense docetaxel followed by doxorubicin and cyclophosphamide with support given as adjuvant or neoadjuvant treatment of women with node positive and high risk breast cancer

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will receive:

Neoadjuvant Docetaxel + Doxorubicin + Cyclophosphamide + Surgery

Adjuvant patients will enter the study after surgery and receive Docetaxel+ Doxorubicin + Cyclophosphamide. Patients treated with lumpectomy will undergo postoperative radiation therapy after completion of chemotherapy. Patients with positive estrogen and/or progesterone receptors will begin anti-estrogen therapy after the last course of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Histologically proven breast cancer
* Females, age greater than 18 years
* Ability to perform activites of daily living with minimal assistance
* Normal cardiac function
* Adequate bone marrow, liver and kidney
* Signed informed consent prior to beginning specific protocol procedures

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Prior systemic anticancer therapy for breast cancer
* Prior anthracycline or taxane based chemotherapy for any malignancy
* Pregnant or breast-feeding women.
* Pre-existing moderate to severe motor or sensory neurotoxicity
* Other serious illness or medical condition

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2004-03; Primary Completion 2005-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Treatment-related toxicities

SECONDARY OUTCOMES:
Overall response rate
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Yardley DA, Burris HA 3rd, Farley CP, Barton JH, Peacock NW, Spigel DR, Greco FA, Hainsworth JD. A phase II feasibility trial of dose-dense docetaxel followed by doxorubicin/cyclophosphamide as adjuvant or neoadjuvant treatment for women with node-positive or high-risk node-negative breast cancer. Clin Breast Cancer. 2008 Jun;8(3):242-8. doi: 10.3816/CBC.2008.n.027. PMID 18650154
- See also: Published article in Clinical Breast Cancer — http://cigjournals.metapress.com/content/a801t38m78tvw61w/fulltext.pdf